CLINICAL TRIAL: NCT05302115
Title: coHOrte fraNcaise Des dEfibrillateurs Sous cuTanés
Brief Title: S-ICD French Cohort Study (HONEST)
Acronym: HONEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paris Sudden Death Expertise Center (Other)
Collaborators: Centre Cardio-Thoracique de Monaco (Unknown); Centre Cardiologique du Nord (Other); Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other); Centre Hospitalier Annecy Genevois (Other); Centre Hospitalier Bretagne Atlantique (Other); Centre Hospitalier William Morey - Chalon sur Saône (Other); Centre Hospitalier du Pays d'Aix (Other); Centre Hospitalier Albi (Unknown); Centre Hospitalier Antibes - Juan Les Pins (Unknown); Centre Hospitalier Argenteuil (Other); Centre Hospitalier Henri Duffaut - Avignon (Other); Centre Hospitalier Auxerre (Unknown); Centre Hospitalier de Bastia (Other); Centre Hospitalier de Bigorre - Tarbes (Unknown); Boulogne sur Mer Hospital Center (Other); Centre Hospitalier de Carcassonne (Unknown); Centre hospitalier de Chambéry (Unknown); Centre Hospitalier of Chartres (Other); Centre Hospitalier de Compiègne (Unknown); Centre Hospitalier de Haguenau (Est France) (Unknown); Centre hospitalier de la Polynésie française - Papeete (Unknown); Centre Hospitalier de La Rochelle (Other); Centre Hospitalier de Lens (Other); Ch Mont de Marsan (Other); Centre Hospitalier de Montauban (Other); Centre Hospitalier de Moulins Yzeure (Other); Centre Hospitalier de PAU (Other); Centre Hospitalier de Perigueux (Other); Centre hospitalier de Perpignan (Other); Centre Hospitalier de Roubaix (Other); Centre Hospitalier de Saint-Brieuc (Other); Centre Hospitalier de Troyes (Other); Centre Hospitalier de Valence (Other); Centre Hospitalier de Valenciennes (Network); Centre Hospitalier Departemental Vendee (Other); Centre Hospitalier le Mans (Other); Centre Hospitalier Eure-Seine (Other); Centre Hospitalier Henri Mondor - Aurillac (Unknown); Centre Hospitalier Intercommunal Castres-Mazamet (Unknown); Centre Hospitalier Jacques Cœur - Bourges (Unknown); Centre Hospitalier Libourne (Unknown); Centre Hospitalier Princesse Grace (Other); Centre Hospitalier Régional d'Orléans (Other); Hôpital NOVO (Other); Centre Hospitalier Rodez (Other); Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other); Central Hospital Saint Quentin (Other Government); Centre Hospitalier Saintonge - Saintes (Unknown); Centre Hospitalier Sud Francilien (Other); Centre Hospitalier Territorial- Nouméa (Unknown); Centre Hospitalier Toulon (Unknown); Centre Hospitalier Universitaire de Saint Etienne (Other); Poissy-Saint Germain Hospital (Other); CHR Mercy - Metz (Unknown); Amiens University Hospital (Other); University Hospital, Angers (Other Government); Centre Hospitalier Universitaire de Besancon (Other); University Hospital, Clermont-Ferrand (Other); University Hospital, Bordeaux (Other); University Hospital, Caen (Other); Centre Hospitalier Universitaire de la Réunion (Other); CHU de Lille (Unknown); University Hospital, Limoges (Other); University Hospital, Montpellier (Other); Central Hospital, Nancy, France (Other); Nantes University Hospital (Other); Poitiers University Hospital (Other); CHU de Rouen - Accueil (Other); University Hospital, Strasbourg, France (Other); University Hospital, Toulouse (Other); CHU de Tours (Unknown); Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier Felix Guyon (Other); University Hospital, Grenoble (Other); Centre Hospitalier Régional et Universitaire de Brest (Other); Centre Hospitalier Universitaire de Nice (Other); CHU de Reims (Other); CHU Rennes - Hopital Pontchaillou (Other); Clinique Alleray Labrouste (Unknown); CMC Ambroise Paré (Other); Clinique Belledonne - Grenoble (Unknown); Clinique Claude Bernard - Metz (Unknown); Clinique du Millenaire (Other); Clinique du Parc - Castelnau le Lez - Montpellier (Unknown); Clinique du Tonkin - Lyon - Villeurbane (Unknown); Clinique Saint-Hilaire (Other); Clinique Les Fontaines - Melun (Unknown); Clinique Louis Pasteur Essey-lès-Nancy (Unknown); Clinique Oreliance - Orléans (Unknown); Clinique Pasteur Toulouse (Other); Clinique Rhône Durance - Avignon (Unknown); Clinique Saint Augustin - Bordeaux (Unknown); Clinique Saint Georges - Nice (Unknown); Clinique Saint Pierre - Perpignan (Unknown); Clinique Saint Vincent - Besancon (Unknown); Clinique Saint-Gatien - Tours (Unknown); Clinique Saint Joseph, Liège (Other); GCS Cardiologie - Bayonne (Unknown); Groupe Hospitalier de Bretagne Sud (Other); Groupe Hospitalier du Havre (Other); Raincy Montfermeil Hospital Group (Network); European Georges Pompidou Hospital (Other); Hopital Antoine Beclere (Other); Bichat Hospital (Other); Centre Hospitalier Universitaire de Nīmes (Other); Hôpital de la Croix-Rousse (Other); Hôpital de la Timone (Other); Henri Mondor University Hospital (Other); Hôpital Marie Lannelongue - Le Plessis Robinson (Unknown); Hôpital Necker-Enfants Malades (Other); University Hospital, Marseille (Other); Hopital Nord Franche-Comte (Other); Hôpital Privé Arnault Tzanck - Mougins - Sophia Antipolis (Unknown); Hôpital privé Bois Bernard - Lens (Unknown); Hôpital privé Clairval - Marseille (Unknown); Hôpital privé Claude Galien - Quincy-sous-Sénart (Unknown); Hôpital Privé de la Loire- Saint Etienne (Unknown); Hôpital Privé de Parly II - Le Chesnay (Other); Hôpital privé du Confluent - Nantes (Unknown); Hôpital privé Le Bois - Lille MetropoleHôpital Privé Les Franciscaines - Nîmes (Unknown); Hôpital Privé Marseille - Beauregard (Unknown); Hôpital privé Saint-Martin - Caen (Unknown); Hospital St. Joseph, Marseille, France (Other); Hôpital Saint Philibert - Lille - GHICL (Unknown); Hospices Civils de Lyon (Other); Institut Jacques Cartier - Massy (Unknown); Institut Mutualiste Montsouris (Other); Pitié-Salpêtrière Hospital (Other); Pôle Santé République (Other); Pôle Santé Sud - Le Mans (Unknown); Polyclinique Les Fleurs - Toulon (Unknown); Polyclinique Lyon-Nord - Rillieux (Unknown); Polyclinique Reims-Bezannes-Courlancy (Unknown); Polyclinique Saint Laurent - Rennes (Unknown); Polyclinique Vauban - Valencienne (Unknown); Amiens SAS (Unknown)
Responsible Party: Sponsor
Other Study IDs: CNIL2217196
Record Dates: First submitted 2020-12-11; First posted 2022-03-31 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Sudden Cardiac Death; Implantable Defibrillator User
Keywords: outcomes; appropriate shock; complications; subcutaneous
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- S-ICD
  Interventions: Device: S-ICD

INTERVENTIONS:
Device: S-ICD — Implantation of an S-ICD

SUMMARY:
Implantable cardioverter-defibrillators have been proven to be effective in the prevention of sudden cardiac death in high-risk patients. However, it is well acknowledged that such a strategy could be optimised, especially through new technologies/devices. Data on the entirely sub-cutaneous implantable cardioverter defibrillator (S-ICD) published so far come from high-volume centers and/or selected populations. The HONEST Cohort -taking the opportunity of a unique scenario with a single manufacturer and remote monitoring system available- aims to collect retrospectively baseline information as well as follow-up of all patients implanted with an S-ICD in France since the first implant in October 13, 2012 until December 31, 2019. An extended prospective yearly follow-up will be carried out since January 1, 2020 until December 31, 2024.

ELIGIBILITY:
Inclusion Criteria:

* All patients who require S-ICD implantation (new or battery replacement)

Exclusion Criteria:

* Refusal of consent

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All S-ICD patients implanted in France since October 13, 2012
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-10-13 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventricular Arrhythmias | Through study completion, an average of 5 years
  Rate of appropriate ICD therapies for ventricular tachycardia / fibrillation
Device-Related Complications | Through study completion, an average of 5 years
  Rate of complications related to ICD including inappropriate therapies, infection, lead or generator dysfunction
Overall and Specific Mortalities | Through study completion, an average of 5 years
  Overall mortality and causes of death

SECONDARY OUTCOMES:
Early Device-Related Complications | 3 months
  Complications occurring within the 3 months following implantation
Late Device-Related Complications | Through study completion, an average of 5 year
  Complications occurring after 3 months following implantation
Stratified Analyses by Sex, Underlying Heart Disease | Through study completion, an average of 5 year
  Primary and secondary outcomes studied by sex and types of heart diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Cardiovascular Research Center (HONEST Investigators), Paris, France

REFERENCES:
- [Derived] Kerkouri F, Eschalier R, Fareh S, Marquie C, Ait Said M, Amara W, Anselme F, Badoz M, Behar N, Bordachar P, El Bouazzaoui R, Champ Rigot L, Chauvin M, Chevalier P, Da Costa A, Defaye P, Deharo JC, Fauchier L, Gandjbakhch E, Gitenay E, Gourraud JB, Guenancia C, de Guillebon M, Guy-Moyat B, Hermida A, Hourdain J, Jacon P, Khattar P, Laredo M, Jesel L, Lellouche N, Leclercq C, Mansourati V, Maury P, Mondoly P, Pasquie JL, Peyrol M, Pierre B, Ploux S, Potelle C, Sadoul N, Sellal JM, Varlet E, Garcia R, Probst V, Boveda S, Marijon E; HONEST Study Investigators. Defibrillation Testing During Implantation of Subcutaneous Implantable Cardioverter Defibrillators. J Am Coll Cardiol. 2025 Jul 8;86(1):32-45. doi: 10.1016/j.jacc.2025.04.048. PMID 40602942
- [Derived] Sousonis V, Jacon P, Kerkouri F, Garcia R, Marquie C, Amara W, Anselme F, Badenco N, Behar N, Belhameche M, Bouzeman A, Fareh S, Guy-Moyat B, Hermida A, Hourdain J, Jesel L, Khattar P, Khoueiry Z, Laurent G, Manenti V, Mechulan A, Menet A, Milhem A, Mondoly P, Ollitrault P, Perrot D, Peyrol M, Pierre B, Sadoul N, Scarlatti D, Taieb J, Vanesson C, Winum P, Probst V, Marijon E, Defaye P, Boveda S; HONEST Study Investigators. S-ICD Implantation Following TV-ICD: Insights Into Patients With Infections and Abandoned Leads: The HONEST Cohort. JACC Clin Electrophysiol. 2025 Sep;11(9):2049-2060. doi: 10.1016/j.jacep.2025.04.020. Epub 2025 Apr 24. PMID 40358574
- [Derived] Waldmann V, Marquie C, Bessiere F, Perrot D, Anselme F, Badenco N, Barra S, Bertaux G, Blangy H, Bordachar P, Boveda S, Chauvin M, Clementy N, Clerici G, Combes N, Defaye P, Deharo JC, Durand P, Duthoit G, Eschalier R, Fauchier L, Garcia R, Geoffroy O, Gitenay E, Gourraud JB, Guenancia C, Iserin L, Jacon P, Jesel-Morel L, Kerkouri F, Klug D, Koutbi L, Labombarda F, Ladouceur M, Laurent G, Leclercq C, Maille B, Maltret A, Massoulie G, Mondoly P, Ninni S, Ollitrault P, Pasquie JL, Pierre B, Pujadas P, Champ-Rigot L, Sacher F, Sadoul N, Schatz A, Winum P, Milliez PU, Probst V, Marijon E. Subcutaneous Implantable Cardioverter-Defibrillators in Patients With Congenital Heart Disease. J Am Coll Cardiol. 2023 Aug 15;82(7):590-599. doi: 10.1016/j.jacc.2023.05.057. PMID 37558371